## INFORMED CONSENT DOCUMENT AGREEMENT TO BE IN A RESEARCH STUDY

# PROSPECTIVE OBSERVATIONAL AND VALIDATION STUDY USING TIMELAPSE MORPHOMETRY MIRI® IMAGING INCUBATOR (TIMMI STUDY)

NAME OF SPONSOR COMPANY: ESCO Medical

PROTOCOL NUMBER: 2016-TiMMI-001

NAME OF PERSON IN CHARGE OF THE RESEARCH STUDY (STUDY DOCTOR/

**INVESTIGATOR):** Matthew VerMilyea, PhD, HCLD/CC

ADDRESS OF STUDY SITE(S):

Ovation Fertility 6500 N. Mopac Expy Building 3 Suite 3102 Austin, Texas 78731

24 Hour-Number Telephone: (512) 610-7474

#### INTRODUCTION

You are being asked to volunteer for a research study. Please take time to read the following information carefully and discuss it with your doctor, friends and family if you wish. You must read and sign this form before you agree to take part in this study. This form will give you more information about this study. Please ask as many questions as you need to before you decide if you want to be in the study. You should not sign this form if you have any questions that have not been answered. Taking part in a research study is entirely voluntary and you can stop being in the study at any time you want to, without any penalty or impact on your medical care or benefits.

The investigator has not been paid by the sponsor (ESCO Medical) to conduct this research study.

#### PURPOSE OF THE STUDY

You are being asked to take part in this research study because you are having in vitro fertilization (IVF) treatment.

During IVF treatment, your embryos are grown in an incubator that supports growth and development.

The purpose of this study is to evaluate the safety and efficacy of the MIRI-TL time-lapse incubator and CultureCoin dish compared to standard big-box incubators and standard culture dishes used for embryo culture.

This research is investigational as the MIRI-TL time-lapse incubator and the CultureCoin dish are not cleared for use by the Food and Drug Administration (FDA) and are experimental.

#### HOW LONG THE STUDY WILL LAST AND HOW MANY PEOPLE WILL BE IN THE STUDY

Women who are 18 years of age and older and undergoing in vitro fertilization at one of the indicated study sites listed above will be asked to participate in the study. 500 participants will be sought in the United States for this study.

#### TO BE IN THIS STUDY

## Subject Responsibilities:

While participating in this research study, you will need to:

- Be willing and able to follow the study directions and procedures
- Tell the study staff about any side effects or problems
- Ask questions as you think of them
- Tell the investigator or the study staff if you change your mind about staying in the study.

#### WHAT WILL HAPPEN DURING THE STUDY

#### **Study Procedures:**

The procedures in this study are designed to follow the standard medical care at each study site for women having IVF treatment (you will sign a separate consent at your clinic for your IVF procedures). Your doctor will explain in detail the procedures you will undergo at your clinic, this form is only meant to explain the details of the research study. This study does include randomization into two different treatment groups, but no sham procedures will be done. A sham procedure is a procedure that has no effect or active treatment.

#### Randomization

Patients will be randomized to the control and study group at the time consent to participate in the study is received. Patients will either be randomized to the MIRI-TL group (MIRI) or the Standard culture group (SC). Randomization means that you will be assigned to a group by chance, like flipping a coin. Neither you, nor your study doctor can choose which group you will be in. You have a 3 in 5 chance of being assigned to the MIRI-TL group and a 2 in 5 chance of being assigned to the Standard Culture group.

## **Embryo Culture Procedures**

Following randomization and standard ovarian stimulation protocols to obtain a sufficient number of mature (MII) oocytes, these oocytes will be fertilized by Intra-Cytoplasmic Sperm Injection (ICSI). If a patient has been randomized to the study group, all inseminated oocytes and subsequently all fertilized diploid (2PN) zygotes will be placed in the CultureCoin and then into the MIRI-TL Time-lapse incubator and cultured as per normal protocol to the blastocyst stage (Day 5/6 or 7). Top quality blastocyst(s) will be transferred and monitored for implantation, pregnancy and ongoing birth. Embryo transfers will either occur in a fresh or frozen embryo transfer cycle.

## **Pregnancy Confirmation (After Embryo Transfer)**

- After embryo transfer, your follow-up visits will take place according to the normal schedule for your clinic and as determined by your doctor.
- About 12-18 days after the egg retrieval, you will have your blood drawn for a standard pregnancy test.
  - o If the result is negative, your participation in the study will be complete.
  - If the test result is positive, you will have an ultrasound examination between 5-8 weeks gestational age to evaluate if a clinical pregnancy has been achieved.
    - If the result is negative, your participation in the study will be complete.
- At between 8-12 weeks gestational age, you will have a second ultrasound examination to verify if your pregnancy is ongoing.
  - o If the result is negative, your participation in the study will be complete.
  - If the test result is positive, you will be followed up until the final outcome of your pregnancy.
- Finally, you will be followed up until your pregnancy concludes with delivery of your baby, or pregnancy termination.
  - o Your study participation will be complete after your pregnancy is concluded.

#### POSSIBLE SIDE EFFECTS AND RISKS

If you do not understand what any of these side effects mean, please ask the investigator or study staff to explain these terms to you.

Potential risks and discomforts associated with the standard medical procedures you may undergo during IVF treatment will be discussed with you by your study doctor. Although those risks are well documented, there may be risks that are not known at this time. IVF may not result in a pregnancy.

## Risks Related to the Study

Potential risks associated with this study are believed to be similar to those related to standard embryo culture protocols. The MIRI-TL and the Culture Coin are CE Marked and have therefore fulfilled European Union (EU) safety and performance criteria. Therefore, both products pose a non-significant risk to participants. The device has been designed with safety specifications and the site will receive training on how to use it prior to the research starting. The device is validated and tested to ensure it is running optimally prior to the start of the research. Compartments are numbered and labelled to avoid errors. However, since the device is investigational, there may be risks that are not yet known.

#### **IVF-Related Risks**

There are discomforts and risks that may be associated with standard medical procedures related to IVF treatment that are not uniquely associated with the use of the study culture media. These risks may include those related to medications, blood draw procedures, egg retrieval, embryo transfer, and follow-up testing.

Other risks may include, but may not be limited to:

- Contamination of the eggs, sperm and/or embryos in the lab.
- Damage to the eggs or embryos during incubation or handling.
- Unforeseen risks such as malfunction of the lab equipment, lab accidents, and/or natural disasters.

You must tell the investigator or study staff about all side effects that you have. If you are not honest about your side effects, it may not be safe for you to stay in the study.

There may be side effects that are not known at this time.

#### POSSIBLE BENEFITS OF THE STUDY

Since this study is for research only, you are not expected to receive any medical benefit. However, the data collected in this study may lead to more effective methods of visualizing, monitoring, culturing and selecting the most viable embryo(s) in order to maximize the chances for implantation and successful pregnancy outcome for future patients.

Subjects in the MIRI-TL group who successfully complete all study procedures will have the option to receive a video of the embryo(s) which was transferred or embryo(s) which were cryopreserved. No reimbursement will be provided for the IVF cycle.

#### **ALTERNATIVES TO PARTICIPATING IN THE STUDY**

Since this study is for research, the only alternative is not to participate. You do not need to be in this study to receive IVF treatment.

#### WITHDRAWL

You can choose to withdraw from the study at any time. If you choose to withdraw your embryos will be removed from the MIRI-TL Time-lapse incubator and placed in the standard incubator used for standard care. If you choose to withdraw, we will ask you if you are willing for us to continue to use the information you have provided for research purposes. You can choose to withdraw any health information you have provided as a participant in the study, at any time and our standard of care will be maintained whether you continue participation or not.

#### CONFIDENTIALITY

Your records of being in this study will be kept private except when ordered by law. The following people will have access to your study records:

The investigator and the research team.

- ESCO Medical, the Sponsor of this study, or those who work for or represent the sponsor
- The United States Food and Drug Administration (FDA)
- Aspire Independent Review Board

A description of this clinical study will be available on <a href="www.ClinicalTrials.gov">www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time. If the study results are presented at meetings or printed in publications, your name will not be used.

#### IN CASE OF STUDY RELATED INJURY

While you are participating in the study you should continue to seek medical advice from you General Practitioner if you believe it is necessary. You can discuss any concerns you have about fertility treatment with your physician. If you have concerns about your participation in the study you can discuss these with the Lead Investigators of each study site. Contact information below.

#### **LEGAL RIGHTS**

You will not lose any of your legal rights by signing this consent form.

#### CONTACT INFORMATION

If you have questions, concerns, or complaints about this study or to report a study related injury, contact:

Matthew VerMilyea, PhD, HCLD/CC Laboratory Director tex@austinIVF.com TEL: (512) 610-7474

If you are unable to reach anyone at the number(s) listed above and you need medical attention, please go to the nearest emergency room.

This study was reviewed by Aspire Independent Review Board (IRB). An IRB reviews research to protect the rights and welfare of study participants. If you have questions, concerns, complaints and/or for information about your rights as a research subject, please call Aspire's Subject Protection Specialist at 1-877-366-5414 (toll free).

Although Aspire IRB has approved the information provided in this informed consent form and has granted approval for the investigator to conduct the study this does not mean Aspire has approved your being part of the study. You need to read the information in this informed consent form for yourself and decide whether or not you want to be in this study.

#### **VOLUNTEERING TO BE IN THE STUDY**

It is your choice if you want to be in the study. No one can force you to be in the study. You may not want to be in this study or you may leave the study at any time without penalty or loss of benefits to which you are otherwise entitled.

The investigator, the sponsor company, or the FDA may take you out of the study without your permission, at any time, for the following reasons:

- If you do not follow the investigator's instructions
- If it is in your best interest;
- You do not consent to continue in the study after being told of changes in the research that may affect you;
- You do not meet all eligibility criteria or you have an embryo transfer before Day 5.
- If the study is stopped

If information generated from this study is published or presented, your identity will not be revealed. If you leave the study, no more information about you will be collected for this study. However, all of the information collected before you left the study will still be used.

#### **ADDITIONAL COSTS**

You will be billed for any standard medical care given during this research study. There will not be any additional costs from taking part in this study. However, you will be responsible for all costs related to your IVF treatments.

#### **NEW FINDINGS**

If there is new information or any significant new findings that could relate to your willingness to continue participation we will tell you. You can then decide if you still want to be in the study.

#### AGREEMENT TO BE IN THE STUDY

I have read this consent form. I understand the purpose, procedures and risks as explained in this document. My questions have been answered to my satisfaction. I voluntarily agree to participate in this study. I know that I can stop participation at any time. I will be given a signed and dated copy of this agreement.

By signing this consent form. I have not given up any of my legal rights.

| by origining and concountrions, related not given up any or my res | ,g |
|---|---|
| Name of Study Subject (printed) | |
| Signature of Study Subject | <br>Date |
| Name of Study Subject's Partner (printed) – if applicable | - |
| Signature of Study Subject's Partner – if applicable | <br>Date |
| Person Obtaining Consent | |
| I have discussed the research study with the subject and subject them in non-technical terms all of the information contained in the including any risks that may reasonably be expected to occur encouraged the subject and the subject's partner to ask questions a were answered. | his informed consent form,<br>r. I further certify that I |
| Printed Name of Person Explaining Consent Form | |
| Signature of Person Explaining Consent Form | <br>Date |
| You will be given a signed and dated copy of this informed consent | to keep. |

#### AUTHORIZATION TO USE AND DISCLOSE INFORMATION FOR RESEARCH PURPOSES

Because information about you and your health is personal and private, it generally cannot be used in this research study without your written authorization. If you sign this form, it will provide that authorization. The form is intended to inform you about how your health information will be used or disclosed in the study. Your information will only be used in accordance with this authorization form and the informed consent form and as required or allowed by law. Please read it carefully before signing it.

## What is the purpose of this research study and how will my health information be utilized in the study?

The purpose of this study is to demonstrate and validate the non-inferior or superior safety and efficacy of the MIRI-TL time-lapse incubator compared to standard big-box incubators used for embryo culture. The procedures in this study are designed to follow the standard medical care for women having in vitro fertilization (IVF).

## Do I have to sign this authorization form?

You do not have to sign this authorization form. But if you do not, you will not be able to participate in this research study.

Signing the form is not a condition for receiving any medical care outside the study.

## If I sign, can I revoke it or withdraw from the research later?

If you decide to participate, you are free to withdraw your authorization regarding the use and disclosure of your health information (and to discontinue any other participation in the study) at any time. After any revocation, your health information will no longer be used or disclosed in the study, except to the extent that the law allows us to continue using your information (e.g., necessary to maintain integrity of research). Information collected before the termination of your authorization may still be used for study purposes. If you wish to revoke your authorization for the research use or disclosure of your health information in this study, you must write to the investigator listed on the first page of this informed consent document. Revoking your authorization and choosing to no longer participate in this study, does not affect your treatment or any other benefits to which you would otherwise be entitled. You will no longer be a part of this research study. The study doctor and staff can continue to share any of the information that they already have.

### What Information Will Be Obtained, Used or Disclosed?

Your health information related to this study, may be used or disclosed in connection with this research study, including, but not limited to, date of birth, ethnicity, fertility history, IVF stimulation protocol, egg retrieval and embryo transfer data, lab results, and clinical ultrasound data (if pregnant).

You have a right to see and copy your information, However, you will not be able to see it while the research study is going on.

## Why will this information be used and/or given to others?

- To do the research.
- To study the results, and
- To see if the research was done correctly

## Who May Use or Disclose the Information?

The following parties are authorized to use and/or disclose your health information in connection with this research study:

- The study investigator and research staff
- The study sponsor
- Aspire Independent Review Board
- The U.S Food and Drug Administration

There may be other information that may be used and given to others that has not been stated above. You should discuss this with the study doctor or a member of the staff and ask any questions that you may have about the sharing of your health information.

## When will my authorization expire?

Your authorization for the use and/or disclosure of your health information will end on December 31, 2020 or when the research project ends, whichever is earlier. I agree to share my information as described in this form and I have received a signed and dated copy for my records.

| Signature of Subject | Date |
|--------------------------------|------|
| , | |
| Signature of Subject's Partner | Date |